CLINICAL TRIAL: NCT04353505
Title: Intra-arterial Sphenopalatine Ganglion Block for Patients With Refractory Headache
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI closed the study before any enrollment
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-11021096
Record Dates: First submitted 2020-03-10; First posted 2020-04-20 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Chronic Migraine; Cluster Headache; Trigeminal Neuralgia
MeSH Terms: conditions — Cluster Headache; Trigeminal Neuralgia | interventions — Ketorolac; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intra-Arterial Delivery of Ketorolac and Dexamethasone (Experimental)
  Interventions: Drug: Ketorolac; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ketorolac — Intra-arterial delivery of Ketorolac in the internal maxillary artery, once
Drug: Dexamethasone — Intra-arterial delivery of Dexamethasone in the internal maxillary artery, once.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of intra-arterial (IA) delivery of Dexamethasone and Ketorolac into the arteries supplying the sphenopalatine ganglion (SPG) - a collection of neurons that plays an important role in headache disorders - in patients with refractory migraine, cluster headache and trigeminal neuralgia. All patients must fail standard treatments prior to enrollment in the trial.

DETAILED DESCRIPTION:
The investigators propose an outpatient, minimally invasive method to deliver Dexamethasone and Ketorolac to the SPG via the intra-arterial route. A microcatheter will be advanced via the radial (preferably) or the femoral artery (in case the radial approach is not feasible) using fluoroscopic guidance and standard interventional techniques, into the distal internal maxillary artery. This artery is a branch of the external carotid artery and supplies the territory of the sphenopalatine ganglion. The microcatheter will be advanced to the ostium of the distal small branches that supply the SPG (i.e. small arteries feeding the vasa nervosum). Once the microcatheter is in a good position, 15 mg Dexamethasone Sodium Phosphate and 15 mg of Ketorolac Tromethamine will be infused over 30 minutes.

The procedure will be performed with local anesthetic at the arterial puncture site. Conscious sedation will be used for anxious participants. After the procedure, the participant will be observed for 5 hours in ICU setting and then discharged to home.

The procedure will be performed unilaterally for participants with cluster headache and trigeminal neuralgia. The procedure could be performed bilaterally for participants with migraine.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of one of the three following headache or facial pain disorders as defined by the ICHD-329 [chronic migraine, cluster headache, trigeminal neuralgia] and failure to respond to two or more preventive therapies

A. Chronic migraine

Failure to respond to two or more preventive therapies including Onabotulinumtoxin A, erenumab, fremanezumab, galcanezumab, topiramate, valproic acid, metoprolol, propranolol, timolol, atenolol, nadolol, amitriptyline, nortriptyline, venlafaxine, duloxetine.

This will include status migrainosus.

B. Cluster headache

Failure to respond to Verapamil, AND one other preventive treatment including Prednisone, Dexamethasone, galcanezumab, lithium, valproic acid, topiramate, external vagus nerve stimulation

C. Trigeminal neuralgia

Failure to respond to two or more preventive therapies, including: Oxcarbazepine or carbamazepine, and One of the following: gabapentin, pregabalin, baclofen, lamotrigine, phenytoin

Exclusion Criteria:

* Patients with malignant neoplasm of the pterygopalatine fossa
* Pregnancy, lactation
* Severe allergic reaction to Dexamethasone
* Severe allergic reaction to NSAID
* Renal failure
* Active systemic infection or fever
* Known cerebral vascular disease
* Drug or alcohol abuse
* Opioid dependency (stable doses ok)
* Triptans within 48 hours from the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Number of Procedure-Related Adverse Events | up to 1 hour post-procedure
Number of Procedure-Related Adverse Events | 5 hours post procedure
Number of Procedure-Related Adverse Events | 2 weeks post procedure

SECONDARY OUTCOMES:
Change in Number of Days of Headache in Subjects with Chronic Migraine | 1 week, 2 weeks, 4 weeks, 6 weeks
Proportion of Chronic Migraine Patients that achieve at least 50% reduction in days of headache frequency | 1 week, 2 weeks, 4 weeks, 6 weeks
Proportion of patients with Cluster Headache that achieve 50% reduction in median number of attacks per day | 1 week, 2 weeks, 4 weeks, 6 weeks
Change in number of days of facial pain for subjects with trigeminal neuralgia | 1 week, 2 weeks, 4 weeks, 6 weeks
Proportion of patients with trigeminal neuralgia that achieve at least 50% reduction in days of facial pain frequency | 1 week, 2 weeks, 4 weeks, 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Athos Patsalides, MD, MPH, Principal Investigator — WCMC
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No